CLINICAL TRIAL: NCT03833596
Title: Synergistic Effect of Exclusive Enteral Nutrition Formula in Addition to Corticosteroids Therapy to Induce Clinical Remission in Patients With Crohn's Disease: a Pilot Study Involving a Multidimensional Assessment of Potential Mechanisms
Brief Title: Exclusive Enteral Nutrition and Corticosteroids Therapy in Crohn's Disease (EENCD)
Acronym: EENCD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: McMaster University (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Maria Ines Pinto Sanchez, Assistant Professor, Department of Medicine, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EEN in Crohn
Record Dates: First submitted 2018-12-21; First posted 2019-02-07 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2019-02

CONDITIONS: Crohn's Disease
Keywords: Corticosteroids; Exclusive Enteral Nutrition
MeSH Terms: conditions — Crohn Disease | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Randomized control trial with three arms of treatment: EEN plus standard or short course of CS versus CS alone.
Masking Description: Treatment options are randomized and masked for participants and study staff until Visit 2, where participants and investigators are made aware of treatment arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard course CS with Regular Food (Active Comparator): 40 mg a day of oral Prednisone for 2 weeks with subsequent taper of daily dose by 5 mg per week.
  Interventions: Drug: Prednisone
- Standard course CS with EEN (Experimental): 40 mg a day of oral Prednisone for 2 weeks and taper of daily dose by 5 mg per week and Exclusive Enteral Nutrition for 6 weeks.
  Interventions: Drug: Prednisone; Dietary Supplement: Exclusive Enteral Nutrition
- Short course CS with EEN (Experimental): 40 mg a day of oral Prednisone for 3 days and taper of daily dose by 5 mg every 3 days and Exclusive Enteral Nutrition for 6 weeks.
  Interventions: Drug: Prednisone; Dietary Supplement: Exclusive Enteral Nutrition

INTERVENTIONS:
Drug: Prednisone — All 3 arms will receive Prednisone - 2 will be standard course treatment, 1 will be short course and rapidly-tapered
Dietary Supplement: Exclusive Enteral Nutrition — 2 arms will receive EEN, in concurrence with either regular-course or short course and rapidly-tapered CS.
  Other Names: Modulen (Nestlé)
  Arms: Short course CS with EEN; Standard course CS with EEN

SUMMARY:
This study evaluates the effect of Exclusive Enteral Nutrition (EEN) in addition to different regimes of corticosteroid (CS) therapy (Prednisone) compared to CS alone in adults participants with active Crohn's Disease, on symptoms and inflammation after 6 weeks of treatment. Participants will be randomized to three treatment arms: standard CS, standard CS with EEN, short course CS with EEN. Participants will be assessed through questionnaires for gut symptoms, quality of life, mood changes and dietary patterns and potential mechanisms will be investigated by collecting stool samples for characterization of gut bacterial profiles, collection of blood to determine inflammatory markers and evaluation of gut motility before and after treatment. The investigators hypothesize that six weeks of EEN with CS will be more effective than CS alone in inducing clinical remission in patients with active CD, as well as leading to beneficial changes in the composition and/or metabolic activity of the intestinal microbiota, gastrointestinal transit and inflammatory burden. Furthermore, six weeks of EEN in addition to a short course of CS will have similar efficacy than EEN with standard course of CS and reduced number of adverse events.

DETAILED DESCRIPTION:
Crohn's disease (CD) is an inflammatory bowel disease (IBD) characterized by diarrhea, abdominal pain and bleeding. There are several treatment options but the most-widely used for acute therapy are corticosteroids (CS), however, CS are often associated with severe side effects. The administration of a formula for exclusive feeding (EEN) is well-established as an alternative to CS in children with Crohn's disease (CD). EEN has been proposed to reduce inflammation in the gut. However, this intervention is not routinely used in adults, in part because of uncertainty regarding the magnitude of the benefit of EEN reported in previous studies. Although few studies have examined the effects of EEN in adult patients with active CD, the potentially synergistic effects of adding EEN to the conventional CS was not explored. Furthermore, it is also possible that the addition of EEN allows to decrease the duration of CS therapy; however, this was not investigated before.

The investigators propose that an oral formula may help decrease gut inflammation and improve nutritional status through modulation of gut bacteria. The investigators will therefore evaluate the effect of exclusive formula feeding therapy in addition to different regimes of CS therapy compared to CS alone in adult patients with active CD, on symptoms and inflammation after 6 weeks of treatment. Participants will be randomized to three treatment arms: standard CS, standard CS with EEN, short course CS with EEN. The investigators will collect information through questionnaires that assess gut symptoms, quality of life, mood changes and dietary patterns. To investigate potential mechanisms, the investigators will collect stool samples to characterize gut bacterial profiles, blood to determine inflammatory markers and evaluate gut movements (motility) before, and after the treatment. The investigators hope that the results will lead to better understanding of the beneficial effect of exclusive formula feeding in addition to CS as a more efficacious alternative than CS alone, and to understand the mechanisms of this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed CD for at least 6 months
* Clinically active disease (CDAI >220 or Harvey-Bradshaw Index (HBI) >6) or active by endoscopy.
* Biochemical evidence of disease activity (CRP >5 and/or fecal calprotectin >250)

Exclusion Criteria:

* Currently using EEN
* Condition that would preclude the use of EEN, such as Intestinal obstruction, perforation, toxic megacolon, massive gastrointestinal bleeding, abdominal abscess, or stricturing disease
* Previous intestinal resection with a remnant bowel of less than 180 cm
* Treatment with Prednisone in the last 30 days
* New start or change in dose of azathioprine, 6-mercaptopurine, cyclosporine, other immunosuppressant or biologics in the last 90 days. Doses of these medications must also remain unchanged for the duration of the study
* New start or change in dose of 5-aminosalicylic acid (ASA) in the last 30 days. 5ASA dose must remain unchanged for the duration of the study
* Use of Antibiotics or Probiotics in the last 30 days
* Pregnant or Lactating
* Any serious illness which could interfere with study procedures or results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of 6 weeks of EEN and CS in inducing remission (Crohn's Disease Activity Index - CDAI<150) in adult patients with active CD (CDAI>220 and either CRP>5 or fecal calprotectin >250mg/l) | 2 years
  Assess the efficacy of 6 weeks of EEN and CS in inducing remission (Crohn's Disease Activity Index (CDAI)<150) compared to treatment with CS alone in adult patients with active CD (CDAI>220 and either CRP>5 or fecal calprotectin >250mg/l)

SECONDARY OUTCOMES:
Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in inducing clinical disease improvement | 2 years
  Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in inducing clinical disease improvement (drop in Crohns Disease Activity Index - CDAI>70)
Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in improving quality of life | 2 years
  Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in improving quality of life (Short Inflammatory Bowel Disease Questionnaire (SIBDQ)) Total score ranges from 10 to 70 (higher values indicate better outcome). Subscales are divided into systemic (score range 2 to 14), social (score range 2 to 14), bowel (score range 3 to 21) and emotional (score range 3 to 21)
Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in inducing biochemical remission | 2 years
  Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in inducing biochemical remission (normalization of either serum CRP (CRP<5) and/or fecal calprotectin (less than 250mg/l)
Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in normalizing colonic transit | 2 years
  Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in normalizing colonic transit (SHAPE) among those with altered transit at baseline. Participants will take one capsule containing 24 markers and have an X-Ray done on day 5. If >20% markers (6 markers or more) are retained it is considered delayed transit.
Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in decreasing anxiety and/or depression scores | 2 years
  Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in decreasing anxiety and/or depression scores (decrease >2 points in Hospital Anxiety and Depression Scale. Total score ranges from 0 to 42, lower values indicating better outcome. Subscale HAD-A (anxiety) and HAD-D (depression) range from 0 to 21.
Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in increasing body weight and improving nutritional status | 2 years
  Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in increasing body weight and improving nutritional status (increased levels of micronutrients: vitamin A, vitamin B12, 25-hydroxy vitamin D, chromium, copper and zinc)
Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in decreasing number of adverse events | 2 years
  Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in decreasing number of adverse events
Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in inducing changes in microbiota composition | 2 years
  Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in inducing changes in microbiota composition (change in alpha diversity by 16S sequencing Illumina)
Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in decreasing indirect markers of mucosal integrity | 2 years
  Determine the beneficial effect of 6 weeks of EEN and CS as compared to CS alone in decreasing indirect markers of mucosal integrity (IFABP2)

CONTACTS AND LOCATIONS:
Overall Officials: Maria I Pinto-Sanchez, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, on, Ontario, Canada

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT03833596/Prot_SAP_000.pdf